CLINICAL TRIAL: NCT05173558
Title: Breaking of Sitting Time Prevents Lower Leg Swelling - Comparison Among Sit, Stand and Intermittent (Sit-to-stand Transitions) Conditions
Brief Title: Breaking of Sitting Time Prevents Lower Leg Swelling
Acronym: Break_sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Analiza Mónica Lopes Almeida Silva, Assistant Professor, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Break_Sitt
Record Dates: First submitted 2021-11-30; First posted 2021-12-30 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Edema Leg
Keywords: Bioimpedance; Raw BIA parameters; Extracellular water expansion; Sedentary behaviour

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Uninterrupted motionless standing (Experimental): 20minutes of uninterrupted motionless standing
  Interventions: Behavioral: Uninterrupted motionless standing
- Uninterrupted motionless sitting (Experimental): 20 minutes of uninterrupted motionless sitting
  Interventions: Behavioral: Uninterrupted motionless sitting
- Sit-to-stand transitions (Experimental): 20 minutes of sit-to-stand transitions (1 minute sitting with 1 minute standing)
  Interventions: Behavioral: Sit-to-stand transitions

INTERVENTIONS:
Behavioral: Uninterrupted motionless standing — Participants remained 20 minutes of uninterrupted motionless standing
  Arms: Uninterrupted motionless standing
Behavioral: Uninterrupted motionless sitting — Participants remained 20 minutes of uninterrupted motionless sitting
  Arms: Uninterrupted motionless sitting
Behavioral: Sit-to-stand transitions — 20 minutes of sit-to-stand transitions (1 minute sitting with 1 minute standing)
  Arms: Sit-to-stand transitions

SUMMARY:
Sitting or standing during a prolonged and uninterrupted period of time is related to negative health outcomes, such as lower extremity swelling. It is unknown if interrupting sedentary behavior by including brief bouts of standing up to the sitting time can attenuate lower leg swelling. Thus, our purpose is to examine if breaking sitting time by adding sit-to-stand transitions attenuates or even prevents lower leg swelling, compared with uninterrupted motionless standing and uninterrupted motionless sitting, using localized bioelectrical impedance raw parameters.

DETAILED DESCRIPTION:
Increased sedentary behavior has deleterious effects on cognitive function, mental health, physical function, disability as well as quality-of-life. Nowadays, prolonged sitting time has been introduced into many situations such as transportation and in the workplace. Staying in the same position (e.g., sitting/standing) for a long and uninterrupted period is associated with poorer health-outcomes, increasing the risk for premature mortality. For instance, sitting for a long period of time has been associated with lower limbs edema. This condition causes discomfort and pain, in turn associated with a lower quality-of-life.

The literature shows that interruption of prolonged sitting time has a positive impact in several health-related risk factors. However, no studies analyzed the effects of motionless sitting with brief standing bouts on lower leg swelling. Thus, the aim of this study is to examine and to compare the effects of standing, sitting and sit-to-stand transitions on lower leg swelling using localized bioelectrical impedance analysis (BIA) measurements A crossover randomized experiment was performed among 20 healthy individuals [age: 27.5±5.9y, 47% females]. In this study, the participants performed the 3 conditions (randomly ordered): 1) uninterrupted motionless standing; 2) uninterrupted motionless sitting; 3) sit-to-stand transitions (1 minute sitting followed by 1 minute standing). Before each condition, a 10-min resting period was performed. Total fat and fat-free mass were determined by dual-energy x-ray absorptiometry. Localized resistance (R), reactance (Xc), impedance (Z) and phase angle (PhA) were assessed at the baseline, at 10 min and at 20 min for each condition.

The researchers hypothesized that interrupting a prolonged sitting position with sit-to-stand transitions will result in greater muscle pump, preventing lower leg swelling.

ELIGIBILITY:
Inclusion Criteria:

* BMI ranging between 18.5 to 29.9 kg/m2;
* Not taking any medications at the time of the measurements;
* All women should have a (self-reported) regular menstrual cycle.

Exclusion Criteria:

* Self-reported inability to stand for 20min without moving the lower limbs
* An active smoking status
* Presence of diabetes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Phase Angle (º) | 8 weeks
  The bioimpedance AKERN BIA 101/BIVA PRO was used to assess physical parameters. Akern is a phase-sensitive device that measures phase angle (PhA).
Impedance (Ohm) | 8 weeks
  The bioimpedance AKERN BIA 101/BIVA PRO was used to assess physical parameters. Akern is a phase-sensitive device that measures impedance (Z).
Resistance (Ohm) | 8 weeks
  The bioimpedance AKERN BIA 101/BIVA PRO was used to assess physical parameters. Akern is a phase-sensitive device that measures phase angle (PhA) and impedance (Z), and then calculates resistance (R).
Reactance (Ohm) | 8 weeks
  The bioimpedance AKERN BIA 101/BIVA PRO was used to assess physical parameters. Akern is a phase-sensitive device that measures phase angle (PhA) and impedance (Z), and then calculates reactance (Xc).

SECONDARY OUTCOMES:
Fat Free Mass (kg) | 8 weeks
  Dual-energy X-ray absorptiometry (DXA; Hologic Explorer-W, Waltham, USA) was used to determine fat-free mass (FFM). A whole-body scan was performed, and the attenuation of X-rays pulsed between 70 and 140kV synchronously with the line frequency for each pixel of the scanned image was measured
Fat mass (kg) | 8 weeks
  Dual-energy X-ray absorptiometry (DXA; Hologic Explorer-W, Waltham, USA) was used to determine total fat mass (FM). A whole-body scan was performed, and the attenuation of X-rays pulsed between 70 and 140kV synchronously with the line frequency for each pixel of the scanned image was measured.
Weight (kg) | 8 weeks
  Weight was measured in bathing suit and no shoes to the nearest 0.01kg using a weight scale.
Height (cm) | 8 weeks
  Height was measured in bathing suit and no shoes to the nearest 0.1cm using a a stadiometer (Seca, Hamburg, Germany), respectively.
Blood pressure (mmHg) | 8 weeks
  Blood pressure was measured (seated and bipedal) right before the start of each protocol. During the experimental condition, blood pressure was measured every 5 minutes.
Heart Rate (bpm) | 8 weeks
  Heart rate was measured (seated and bipedal) right before the start of each protocol. During the experimental condition, heart rate was measured every 5 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Motricidade Humana, Oeiras, Cruz-Quebrada, Portugal

IPD SHARING:
Plan to Share IPD: No